CLINICAL TRIAL: NCT01558349
Title: Circulating Tumor Cells and Melanoma: Comparing the EPISPOT (EPithelial ImmunoSPOT) and CellSearch Techniques
Brief Title: Circulating Tumor Cells and Melanoma: Comparing the EPISPOT and CellSearch Techniques
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2011/LM-05; 2012-A00236-37 (Other: ANSM)
Record Dates: First submitted 2012-03-17; First posted 2012-03-20 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2017-01

CONDITIONS: Metastatic Melanoma
Keywords: Epispot; CellSearch; Circulating melanoma cells; circulating cells
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hospitalized controls: Patients that have been hospitalized at the Nîmes University Hospital and who do not have dermatological cancer.
- Metastatic melanoma: This cohort includes patients with metastatic melanoma.

SUMMARY:
The main objective of this study is to compare results for the detection of circulating melanoma cells (CMC) using CellSearch versus EPISPOT (EPithelial ImmunoSPOT) techniques between a group of patients with metastatic melanoma and a group of hospitalized control patients.

DETAILED DESCRIPTION:
The secondary objectives of this study include:

A. To compare the following elements between the two patient groups:

* the number of CMCs per ml of blood as determined by EPISPOT
* the number of CMCs per ml of blood as determined by CellSearch
* the percentage of patients with at least 2 CMCs per ml of blood according to the two techniques
* the % of CMCs expressing KI67
* the % of CMCs expressions S100 (only the EPISPOT technique)

B. To compare the EPISPOT and CellSearch techniques is terms of the following:

* the number of CMCs detected per ml blood
* the number of CMCs expressing antigen KI67

C. To re-evaluate the 2-CMC per ml blood threshold

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available, within the hours of his/her normally scheduled medical care, for blood sampling at 8 am and 4 pm on the same day.

Inclusion Criteria for patients:

* Stage 4 melanoma, without other associated neoplasms

Inclusion Criteria for controls:

* Patient without cancer, nor history of cancer

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a contra-indication for a treatment used in this study

Exclusion criteria for patients:

* Stage 1 to 3 melanoma, or other types of cancer

Exclusion criteria for controls:

* History of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The two cohorts in this study are composed of (1) patients suffering from metastatic melanome and (2) hospitalized patients with no history of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2013-06-27 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Presence/absence of at least 2 CMCs per ml blood, both techniques | Day 1 at 8 am
  Presence/absence of at least 2 CMCs per ml blood, using both the Epispot and the CellSearch techniques

SECONDARY OUTCOMES:
CMCs per ml blood, Epispot | Day 1 at 8 am
  The number of CMCs per ml blood as determined by the Epispot technique
CMCs per ml blood, CellSearch | Day 1 at 8 am
  The number of CMCs per ml blood as determined by the CellSearch technique
delta CMC | Day 1 at 8 am
  The difference between the number of CMCs per ml blood detected with the CellSearch technique and the Epispot Technique (CellSearch - Epispot)
% delta CMC | Day 1 at 8 am
  The % difference between the number of CMCs per ml blood detected with the CellSearch technique and the Epispot Technique (CellSearch - Epispot)/CellSearch*100
Presence/absence of KI67 antigen markers | Day 1 at 8 am
% cells with S100 protein markers | Day 1 at 8 am

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Meunier, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Cayrefourcq L, De Roeck A, Garcia C, Stoebner PE, Fichel F, Garima F, Perriard F, Daures JP, Meunier L, Alix-Panabieres C. S100-EPISPOT: A New Tool to Detect Viable Circulating Melanoma Cells. Cells. 2019 Jul 20;8(7):755. doi: 10.3390/cells8070755. PMID 31330795